CLINICAL TRIAL: NCT04525339
Title: Early Outcomes of Concomitant Transcatheter Aortic Valve Implantation and Off-pump Coronary Artery Bypass Grafting in Management of Severe Symptomatic Aortic Stenosis and Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Moustafa Mohamed, Assistant Lecturer of Cardiothoracic Surgery/ Principle Investigator, Assiut University
Other Study IDs: TAVI & OPCAB
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Aortic Valve Disease; Coronary Artery Disease
MeSH Terms: conditions — Aortic Valve Disease; Coronary Artery Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TAVI and Off pump CABG — Concomitant Transcatheter aortic valve implanatation and off pump coronary artery bypass grafting

SUMMARY:
Study Objectives/Specific Aims Overall Goal: To study the outcomes of patients undergoing TAVI, their subsequent results and complications.

* Objective 1: Identify risk factors that are predictive of the need for TAVI and CABG
* Objective3:Assess early 3 months outcomes and postoperative results

Outcome Measure:

1. All-cause mortality within 3 months.

Secondary Outcome Measures:

1. Stroke
2. Myocardial infarction
3. Bleeding
4. Hospital stay
5. Acute kidney injury
6. Number of patients with conduction disturbance and pacemaker implantation
7. Gradient on implanted valve
8. Degree of transvalvular leakage
9. 6 weeks follow-up
10. 3 months Echo

DETAILED DESCRIPTION:
Severe symptomatic aortic stenosis in elderly patients represents a surgical challenge for cardiac surgeons due to heavy calcifications and associated comorbidities. Such conditions usually are associated with dramatic intra and postoperative complications leading to many cases being declined for open surgical replacement. Many treatment modalities were described including trans-catheter valvutomy but with only temporary improvements and high rates of recurrence. Transcatheter Aortic Valve Implantation (TAVI) has offered an alternative solution to such cases in which open surgery is deemed too risky or prohibited.

Coronary artery disease (CAD) is a common comorbidity in patients undergoing TAVI. It has been reported with 40-75% of the patients with increased adverse outcomes.Despite performing TAVI alone in these patient has shown significant improvement, yet CAD has showed increased risk in terms of hemodynamic instability and risk of myocardial infarction during rapid pacing which is an important step during the TAVI procedure.

According to the AHA/ACC guidelines, in patients undergoing Aortic valve replacement/ repair (AVR) who also have significant CAD, the combination of Coronary artery bypass grafting (CABG) and AVR reduces the rates of perioperative Myocardial Infarction, perioperative mortality, late mortality, and morbidity when compared with patients not undergoing simultaneous CABG, even though the combined operation carries a small but real increased risk of mortality (Class II A).

Percutaneous coronary intervention (PCI) has been the commonly used treatment modality for (CAD) which is usually carried out pre TAVI or less commonly simultaneously with TAVI (mainly due to access limitation after valve implantation). In patients with intermediate or high SYNTAX scores, CABG remains the standard therapy. Off-pump coronary artery bypass (OPCAB) procedure has demonstrated excellent results in these patients, due to the avoidance of cardiopulmonary bypass and manipulation of the aorta.

Only a few studies in the literature have reported the combined approach of CABG and TAVI in treatment of coronary artery disease and severe symptomatic aortic stenosis. Here the invesigators decided to study the early three months outcomes of patients undergoing TAVI and surgical revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe symptomatic aortic stenosis and CAD undergoing TAVI & OPCABG

Exclusion Criteria:

* Patients with concomitant valvular heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in cardiac surgery department, Manchester Royal Infirnary in the last five years 2015 till 2020, and who meet the listed inclusion and exclusion criteria will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 months

SECONDARY OUTCOMES:
Occurence of Stroke | I month
Occurence of Myocardial infarction | I month
Need for reexploration | I month
Occurence of Acute kidney injury | I month
Number of patients with conduction disturbance and pacemaker implantation | I month
Gradient on implanted valve | 3 months Echo
Degree of transvalvular leakage | 3 months Echo
Days of Hospital Stay | from day of operation till medically fit for discharge (1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt